CLINICAL TRIAL: NCT04745403
Title: Safety and Tolerability Study of Redirected HBV-Specific T Cells in Patients With Hepatitis B Virus (HBV)-Related Hepatocellular Carcinoma (SAFE-T-HBV)
Brief Title: Redirected HBV-Specific T Cells in Patients With HBV-related HCC (SAFE-T-HBV)
Acronym: SAFE-T-HBV
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lion TCR Pte. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTCR-HCC-3-3
Record Dates: First submitted 2021-01-25; First posted 2021-02-09 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatitis B virus; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mRNA HBV/TCR T-cells (Experimental): Escalating regime from 1x10e5 to 5-10x10e6 cells/kg bodyweight (BW) every 2 weeks.
  Interventions: Drug: mRNA HBV/TCR T-cells

INTERVENTIONS:
Drug: mRNA HBV/TCR T-cells — Study Infusion
  The first dose of mRNA HBV-TCR T-cells at dose 1x10e5/kg BW will be infused on Day 0, and subsequently incremental doses on Day 14 and 28, up to the dose of 5-10x10e6/kg BW.

SUMMARY:
This is a single center, single arm and open-label study to determine the safety of mRNA modified HBV-TCR redirected T-cells and to analyze the changes in tumor microenvironment caused by these HBV-TCR redirected T-cells in subjects with HBV-related HCC who are not amenable to/failed conventional treatment.

ELIGIBILITY:
Key Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status ≤1
2. Presence of primary hepatocellular carcinoma in the liver with presence of measurable tumour by RECIST 1.1 criteria, that is not amenable to, or failed, conventional treatment options
3. Serum HBsAg positivity
4. Non-cirrhotic or compensated cirrhosis Child-Pugh A (5 - 6 points)
5. Life expectancy of at least 3 months
6. HLA class 1 profile matching HLA-class I restriction element of the available T cell receptors (restricted by either HLA-A*02:01 or HLA-A*24:02).

Key Exclusion Criteria:

1. Brain metastasis
2. Second primary malignancy that is clinically detectable at the time of consideration for study enrolment, except for in situ carcinoma of the cervix, non-melanoma skin carcinoma localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer and superficial bladder tumors
3. Use of immune checkpoint inhibitors and/or tyrosine kinase inhibitor (TKI) within 5 half-lives of the drug prior to baseline liver biopsy procedure
4. Alterations of concomitant medications which could potentially cause drug induced liver injury and affect liver biopsy result within 3 months of baseline liver biopsy procedure.
5. Likelihood to require any immunosuppressive treatments during the period of the clinical trial.
6. 7. Last RFA/TACE treatment within 3 months prior to first LioCyx-M infusion; Last Y90 therapy treatment within 6 months prior to first dose of mRNA HBV/TCR T-cells
7. Decompensated cirrhosis Child-Pugh B or C (7 - 15 points)
8. Concurrent administration of any other anti-tumour therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
9. Use of any investigational product (IP) or investigational medical device within 30 days of study drug administration
10. Serum HBV DNA levels ≥ 200 IU/ml at screening
11. Serum HBsAg levels ≥ 10,000 IU/ml at screening
12. Lack of peripheral venous or central venous access or any condition that would interfere with drug administration or collection of study samples
13. Any condition or active infections which, in the investigator's opinion, makes the subject unsuitable for trial participation
14. Women who are pregnant or breast-feeding

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation of mRNA HBV/TCR T-cell treatment | Start of treatment until 28 days post last dose
  Based on incidence and severity of adverse events
Analysis of modifications of tumour microenvironment caused by mRNA HBV/TCR T-cell treatment | Start of treatment until end of study
  Histological staining using biopsy and analysis of serum factors such as cytokines and chemokines

SECONDARY OUTCOMES:
Evaluation of anti-tumor efficacy of mRNA HBV/TCR T-cell treatment | Up to 4 years
  Objective response rate (ORR)
Evaluation of anti-tumor efficacy of mRNA HBV/TCR T-cell treatment | Up to 4 years
  Progression free survival (PFS)
Evaluation of anti-tumor efficacy of mRNA HBV/TCR T-cell treatment | Up to 4 years
  Overall survival (OS)

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koh S, Shimasaki N, Suwanarusk R, Ho ZZ, Chia A, Banu N, Howland SW, Ong AS, Gehring AJ, Stauss H, Renia L, Sallberg M, Campana D, Bertoletti A. A practical approach to immunotherapy of hepatocellular carcinoma using T cells redirected against hepatitis B virus. Mol Ther Nucleic Acids. 2013 Aug 13;2(8):e114. doi: 10.1038/mtna.2013.43. PMID 23941866
- [Result] Kah J, Koh S, Volz T, Ceccarello E, Allweiss L, Lutgehetmann M, Bertoletti A, Dandri M. Lymphocytes transiently expressing virus-specific T cell receptors reduce hepatitis B virus infection. J Clin Invest. 2017 Aug 1;127(8):3177-3188. doi: 10.1172/JCI93024. Epub 2017 Jul 24. PMID 28737510
- [Result] Tan AT, Yang N, Lee Krishnamoorthy T, Oei V, Chua A, Zhao X, Tan HS, Chia A, Le Bert N, Low D, Tan HK, Kumar R, Irani FG, Ho ZZ, Zhang Q, Guccione E, Wai LE, Koh S, Hwang W, Chow WC, Bertoletti A. Use of Expression Profiles of HBV-DNA Integrated Into Genomes of Hepatocellular Carcinoma Cells to Select T Cells for Immunotherapy. Gastroenterology. 2019 May;156(6):1862-1876.e9. doi: 10.1053/j.gastro.2019.01.251. Epub 2019 Jan 31. PMID 30711630